CLINICAL TRIAL: NCT02336932
Title: Vitamin D and the Free Hormone Hypothesis: Lessons From Surgical Stress
Brief Title: Vitamin D and the Free Hormone Hypothesis
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Martin Blomberg Jensen, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: VITD201501
Record Dates: First submitted 2014-11-13; First posted 2015-01-13 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Arthrosis; Surgery
Keywords: vitamin d; free hormone; surgical stress
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe changes in vitamin D parameters before, during and after a well-defined elective surgical trauma (knee arthroplasty) and to compare these changes to other steroid hormones (testosterone and oestrogens). The hypothesis is that profound changes in free and total vitamin D will occur as a result of changes between intravascular vs extravascular protein compartments during surgical trauma.

DETAILED DESCRIPTION:
Introduction:

Vitamin D is a versatile signaling molecule with a well-established role in the regulation of calcium homeostasis and bone health. The spectrum of vitamin D target-organs has expanded and it has been suggested that vitamin D influences the immune system, endocrine organs such as pancreas, testis and ovary and multiple other organs (Blomberg Jensen 2014). More recently attention has been paid to surgical patients suggesting hypovitaminosis D to increase postoperative morbidity. (Turan A et al, Zaloga et al). However, the perioperative literature is hindered by a mixture of acute and chronic diseases indicating surgery, different types of surgery and different time of vitamin-D assessments (pre- vs post-operatively) (Turan A et al Zaloga et al).

Vitamin-D is a protein-bound steroid hormone and interpretation of vitamin-D surgical studies require knowledge about the effect of clinical surgical trauma per se on vitamin-D physiology, as has been demonstrated with cortisol, thyroid hormones and other steroid hormones (Kehlet, Brandt, Rem). Unlike other steroid hormones vitamin D depends on a two step activation process before it is able to bind and activate the vitamin D receptor (VDR). First by 25-hydroxylation (CYP2R1) in the liver, which forms 25-hydroxyvitamin D (25-OHD). 25-OHD is also biologically inactive but used clinically to determine vitamin D status because serum 25-OHD levels are associated with rickets, bone health and calcium homeostasis. Circulating 25-OHD is bound to vitamin D binding protein (DBP) (Prosser and jones 2004). This complex is filtered in the glomerulus and subsequently transported into the proximal tubules cells by megalin-mediated uptake (Nykjær 1999). Here, 25-OHD undergoes 1α-hydroxylation (CYP27B1) and the resulting 1,25(OH)2D3 binds and activates the vitamin D receptor (VDR). The fact that the protein bound fraction is taken up by megalin differs from the metabolic clearance and/or activation of other steroid hormones and questions whether the free hormone hypothesis is applicable to the vitamin D system. The fact that binding proteins are lost during surgical stress indicates that this patient group is ideal for studying total versus free hormone concentrations and possible secondary changes for instance in serum PTH and calcium due to functional hormonal aberrations.

Aim of study:

The purpose of this study is to describe changes in vitamin D parameters before, during and after a well-defined elective surgical trauma (knee arthroplasty) and to compare these changes to another steroid hormone (testosterone and oestrogens). The hypothesis is that profound changes in free and total vitamin D will occur as a result of changes between intravascular vs extravascular protein compartments during surgical trauma.

DESIGN This is a prospective observational study

Patients and methods 20 otherwise healthy patients (10 males and 10 females) age 50-75 years undergoing elective total knee arthroplasty in Department of Orthopaedic Surgery, Hvidovre Hospital. All patients undergo standard anesthesia and analgesic treatment in a fast-track set-up with discharge not earlier than 48-hours postoperatively.(Husted et al 2011) Exclusion criteria are

* intake of high dose vitamin D (above 10 microgram daily),
* serious co-morbidities such as previous Myocardial Infarction, heart, kidney or liver failure, severe rheumatological disorders, existing endocrine disorders in thyroid, pancreas, testis, adrenal,
* Disorders related to calcium metabolism, hypercalcemia,
* Granulomatous disease such as Wegener, tuberculosis, etc,
* Previous or present malignant disease, inflammatory bowel disease
* Current use of medication that influence protein binding and renal excretion (allopurinol, diuretics, hormones. immunosuppressive therapy)
* Elevated serum creatinine
* Non-european ethnicity

SAMPLE SIZE CALCULATION AND STATISTICS In this association study with 20 participants we estimate based on the studies conducted with cortisol and other steroid hormones that the cohort size is sufficient to show the kinetics in vitamin D metabolism after surgery

SCREENING AND TIME COURSE Men and women, who are investigated at Department of Orthopedics at Hvidovre hospital will be screened for eligibility to the study. Those who meet the criteria for participation will be informed, and if they consent allocated to the study. The study will be initiated January 2015 and ends when the last person has been included latest April 2015.

Each person will have one blood sampling performed prior to surgery and 2, 6, 24 and 48 hours postoperatively. Three weeks after inclusion the patients will have a final blood sample drawn .

Blood samples Venus blood is drawn preoperatively before i.v. fluid administration, 2, 6, 24,48 hours and 3 weeks postoperatively. Serum has to be frozen within 1 hour and will be stored at minus 20 degrees celsius until analysis.

OUTCOME MEASUREMENTS

* Primary endpoints

  •Changes in total and calculated free 25-hydroxyvitamin D and 1,25dihydroxyvitamin D postoperatively.
* Secondary endpoints

  * Serum concentrations of total calcium, albumin corrected calcium, phosphate, alkaline phosphatase, vitamin D binding protein and Parathyroid hormone (PTH)
  * Total and calculated free testosterone and estradiol in males and females respectively.
  * are the changes in sex hormones different from vitamin D
  * Serum gonadotopin levels
  * sex dependence. Are the changes in vitamin D availability dependent on sex.
  * dependence on preoperative vitamin D status. Are the changes in vitamin D availability dependent on baseline serum vitamin D status
  * Changes in serum concentrations of putative regulators and downstream signals osteocalcin, fibroblas growth factor 23 (FGF23), osteopontin, RANKL, osteoprotegerin (OPG), alpha Klotho, Sclerostin and IGF-1.
  * Temporal changes in serum level of binding proteins. differences for vitamin D binding protein, albumin and sex hormone binding globulin.

ANALYSIS AND INTERVENTION

Reproductive hormones and growth factors will be analysed at dept. of GR, Rigshospitalet. Other serum analyses will be analysed at Department of clinical biochemistry, Holbæk and Aarhus Kommune Hospital

ETHICS AND SIDE EFFECTS All the patients will have full-filled their investigation, before they are invited to the study. They will be informed of potential adverse effects, and they can leave the trial at any point without any consequences. All participants will be informed and counselling according to their VD status 3 weeks after the surgery. This study poses no additional risk to the patients except for the 5 perioperative blood samples (each 8 ml in total 40 ml per patient), as everything else is according to standard clinical practice.

PUBLICATION OF RESULTS All results, positive or negative will be submitted to peer reviewed scientific journals. Data will successively be obtained and transferred to a statistical database.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients (10 males and 10 females)
* age 50-75 years
* undergoing elective total knee arthroplasty at Department of Orthopaedic Surgery, Hvidovre Hospital

Exclusion Criteria:

* intake of high dose vitamin D (above 10 microgram daily),
* serious co-morbidities such as previous myocardial infarct, heart, kidney or liver failure, severe rheumatological disorders, existing endocrine disorders in thyroid, pancreas, testis, adrenal,
* Disorders related to calcium metabolism, hypercalcemia,
* Granulomatous disease such as Wegener, tuberculosis, etc,
* Previous or present malignant disease, inflammatory bowel disease
* Current use of medication that influence protein binding and renal excretion (allopurinol, diuretics, hormones. immunosuppressive therapy)
* Elevated serum creatinine
* Non-european ethnicity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 otherwise healthy patients (10 males and 10 females) age 50-75 years undergoing elective total knee arthroplasty in Department of Orthopaedic Surgery, Hvidovre Hospital. All patients undergo standard anaesthesia and analgesic treatment in a fast-track set-up with discharge not earlier than 48-hours postoperatively.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
• Changes in total and calculated free 25-hydroxyvitamin D and 1,25dihydroxyvitamin D postoperatively. | 2, 6, 24,48 hours and 3 weeks postoperatively.
  Changes in serum concentration of total and free vitamin D metabolites

SECONDARY OUTCOMES:
changes in serum concentrations of total calcium, albumin corrected calcium, phosphate, alkaline phosphatase and PTH | 2, 6, 24,48 hours and 3 weeks postoperatively.
•Dependence of sex in the changes in total and calculated free 25-hydroxyvitamin D and 1,25dihydroxyvitamin D, calcium, AP and PTH | 2, 6, 24,48 hours and 3 weeks postoperatively.
  AP alkaline phospatase
• Changes in total and calculated free 25-hydroxyvitamin D and 1,25dihydroxyvitamin D dependent on preoperative vitamin D status | 2, 6, 24,48 hours and 3 weeks postoperatively.
• Secondary changes in serum of FGF23, Klotho, RANKL, OPG, osteocalcin, osteopontin, Sclerostin and IGF-1 | 2, 6, 24,48 hours and 3 weeks postoperatively.
• Temporal changes in serum level of vitamin D binding protein, albumin and sex hormone binding globulin. | 2, 6, 24,48 hours and 3 weeks postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: martin B Jensen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet/Hvidovre hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Blomberg Jensen M. Vitamin D and male reproduction. Nat Rev Endocrinol. 2014 Mar;10(3):175-86. doi: 10.1038/nrendo.2013.262. Epub 2014 Jan 14. PMID 24419359
- [Background] Prosser DE, Jones G. Enzymes involved in the activation and inactivation of vitamin D. Trends Biochem Sci. 2004 Dec;29(12):664-73. doi: 10.1016/j.tibs.2004.10.005. PMID 15544953
- [Background] Nykjaer A, Dragun D, Walther D, Vorum H, Jacobsen C, Herz J, Melsen F, Christensen EI, Willnow TE. An endocytic pathway essential for renal uptake and activation of the steroid 25-(OH) vitamin D3. Cell. 1999 Feb 19;96(4):507-15. doi: 10.1016/s0092-8674(00)80655-8. PMID 10052453
- [Background] Husted H, Lunn TH, Troelsen A, Gaarn-Larsen L, Kristensen BB, Kehlet H. Why still in hospital after fast-track hip and knee arthroplasty? Acta Orthop. 2011 Dec;82(6):679-84. doi: 10.3109/17453674.2011.636682. Epub 2011 Nov 9. PMID 22066560
- [Background] Rem J, Nielsen OS, Brandt MR, Kehlet H. Release mechanisms of postoperative changes in various acute phase proteins and immunoglobulins. Acta Chir Scand Suppl. 1980;502:51-6. PMID 6941601
- [Background] Brandt MR, Kehlet H, Skovsted L, Hansen JM. Rapid decrease in plasma-triiodothyronine during surgery and epidural analgesia independent of afferent neurogenic stimuli and of cortisol. Lancet. 1976 Dec 18;2(7999):1333-6. doi: 10.1016/s0140-6736(76)91977-2. PMID 63806
- [Background] Turan A, Hesler BD, You J, Saager L, Grady M, Komatsu R, Kurz A, Sessler DI. The association of serum vitamin D concentration with serious complications after noncardiac surgery. Anesth Analg. 2014 Sep;119(3):603-612. doi: 10.1213/ANE.0000000000000096. PMID 25121616
- [Background] Zaloga GP, Butterworth JF 4th. Hypovitaminosis D in hospitalized patients: a marker of frailty or a disease requiring treatment? Anesth Analg. 2014 Sep;119(3):613-618. doi: 10.1213/ANE.0000000000000368. No abstract available. PMID 25136999
- [Background] Kehlet H, Madsen SN, Binder C. Cortisol and cortisone acetate in parenteral glucocorticoid therapy? Acta Med Scand. 1974 May;195(5):421-3. doi: 10.1111/j.0954-6820.1974.tb08163.x. No abstract available. PMID 4830060
- [Background] Reid D, Toole BJ, Knox S, Talwar D, Harten J, O'Reilly DS, Blackwell S, Kinsella J, McMillan DC, Wallace AM. The relation between acute changes in the systemic inflammatory response and plasma 25-hydroxyvitamin D concentrations after elective knee arthroplasty. Am J Clin Nutr. 2011 May;93(5):1006-11. doi: 10.3945/ajcn.110.008490. Epub 2011 Mar 16. PMID 21411617
- [Background] Bogunovic L, Kim AD, Beamer BS, Nguyen J, Lane JM. Hypovitaminosis D in patients scheduled to undergo orthopaedic surgery: a single-center analysis. J Bone Joint Surg Am. 2010 Oct 6;92(13):2300-4. doi: 10.2106/JBJS.I.01231. PMID 20926724